CLINICAL TRIAL: NCT00141414
Title: Pregabablin Open-Label, Follow-On Safety Trial In Patients With Refractory Partial Epilepsy.
Brief Title: To Evaluate the Long-Term Safety of Pregabalin in Refractory Partial Epilepsy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1008-008
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2007-01-01 (Estimated); Status verified 2006-12

CONDITIONS: Epilepsy, Partial
MeSH Terms: conditions — Epilepsies, Partial | interventions — Pregabalin

INTERVENTIONS:
Drug: Pregabalin

SUMMARY:
To evaluate the long-term safety of pregabalin in refractory partial epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Must have met the inclusion criteria for preceding double-blind study.
* Have received double-blind study medication and wish to receive open-label pregabalin.

Exclusion Criteria:

* Pregnant or considering becoming pregnant.
* Receiving any concomitant medication that could alter the effectiveness of their medication response or seizure frequency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82
Dates: Start 1997-11; Study Completion 2005-10

PRIMARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- United States (20):
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Stanford, California
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Saint Paul, Minnesota
  - Pfizer Investigational Site, Chesterfield, Missouri
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Madison, Wisconsin
- Pfizer Investigational Site, Bonn, Germany